CLINICAL TRIAL: NCT03155958
Title: Ocular Comorbidities of Alopecia Areata
Brief Title: Ocular Finding in Alopecia Areata
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Walaa Mahmoud, principle investigator, Assiut University
Other Study IDs: OCCAA
Record Dates: First submitted 2017-05-15; First posted 2017-05-16 (Actual); Last update posted 2017-05-16 (Actual); Status verified 2017-05

CONDITIONS: Hair Loss
MeSH Terms: conditions — Alopecia

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Alopecia areata (AA) is a common, idiopathic and sometimes recurrent non-scarring type of hair loss.

Several etiological factors, including psychological, trauma-related, genetic and autoimmune factors have been considered as possible etiological factors . A T cell-mediated autoimmune mechanism in genetically vulnerable individuals is the most acceptable etiology.

Alopecia areata presents clinically with well demarcated patches of non cicatricial hair loss in any hair bearing area with no remarkable gender preference.

Although AA may occur at any age, incidence is high among younger age groups. In fact, it is the most common form of alopecia seen in children. Various clinical patterns of alopecia have been described as patchy, diffuse, reticulate, ophiasis and ophiasis inversus. Depending on the extent of hair loss, it can be classified into alopecia subtotalis, alopecia totalis (complete loss of scalp hair), and alopecia universalis (complete loss of body hair).

National Alopecia Areata Foundation has devised "Severity of Alopecia Tool Score" (SALT score) as a measure of disease severity. Scalp is divided into 4 areas, namely, Vertex-40% of scalp surface area; right and left profiles-18% each and posterior scalp aspect-24%. SALT score is the sum of percentage of hair loss in the above mentioned areas.

DETAILED DESCRIPTION:
Alopecia areata is now considered a systemic autoimmune disease that may have other serious comorbidities, such as cardiovascular and ocular. However, the results of studies of ocular findings in AA are controversial.

Several ocular alterations have been previously reported in patients with AA ranging from minor punctate opacities to cataract. However, there are contrasting opinions on the significance of these lenticular changes. In addition, Horner syndrome, pupil ectopia, iris atrophy, fundus changes , bilateral keratoconus, iris changes and retinal changes have been reported in AA.

Dermoscopy is a noninvasive, diagnostic tool which visualizes subtle patterns of skin lesions not normally visible to the unaided eye. Characteristic dermoscopic finding of AA included black dots , tapering hair corresponding to " exclamation mark hairs " , broken hairs , yellow dots , and clustered short vellus hairs ( shorter than 10 mm).

Since ocular affection can be a profound morbidity factor in patients with AA, we will search deeply in this study about this correlation in order to conclude the value of ocular screening in each and every patient with AA.

ELIGIBILITY:
Inclusion Criteria:

* patients of alopecia areata will be recruited from the Dermatology Outpatients' Clinic, Assiut University Hospitals, Assiut, Egypt.

Exclusion Criteria:

1. Patients with documented eye disease.
2. Patients with any systemic illness.
3. Patients who received any systemic treatment with possible ocular implications in the last three months.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Study subjects will be recruited from the Dermatology Outpatients' Clinic, Assiut University Hospitals, Assiut, Egypt.
Sampling Method: Non-Probability Sample
Enrollment: 1 (Estimated)
Dates: Start 2017-07-01 (Estimated); Primary Completion 2019-07-01 (Estimated); Study Completion 2020-01-01 (Estimated)

PRIMARY OUTCOMES:
the number of patient with occular affection in alopecia areata | 2 years
  percentage

SECONDARY OUTCOMES:
correlate dermoscopic finding with disease severity and ocular finding | 2 years

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Madani S, Shapiro J. Alopecia areata update. J Am Acad Dermatol. 2000 Apr;42(4):549-66; quiz 567-70. PMID 10727299
- [Background] Esmer O, Karadag R, Cakici O, Bilgili SG, Demircan YT, Bayramlar H, Karadag AS. Ocular findings in patients with alopecia areata. Int J Dermatol. 2016 Jul;55(7):814-8. doi: 10.1111/ijd.13114. Epub 2016 Apr 7. PMID 27061214
- [Background] Ergin C, Acar M, Kaya Akis H, Gonul M, Gurdal C. Ocular findings in alopecia areata. Int J Dermatol. 2015 Nov;54(11):1315-8. doi: 10.1111/ijd.12897. Epub 2015 Jul 3. PMID 26147700
- [Background] Price VH. Double-blind, placebo-controlled evaluation of topical minoxidil in extensive alopecia areata. J Am Acad Dermatol. 1987 Mar;16(3 Pt 2):730-6. doi: 10.1016/s0190-9622(87)70095-4. PMID 3549809
- [Background] Pandhi D, Singal A, Gupta R, Das G. Ocular alterations in patients of alopecia areata. J Dermatol. 2009 May;36(5):262-8. doi: 10.1111/j.1346-8138.2009.00636.x. PMID 19382996
- [Background] Recupero SM, Abdolrahimzadeh S, De Dominicis M, Mollo R, Carboni I, Rota L, Calvieri S. Ocular alterations in alopecia areata. Eye (Lond). 1999 Oct;13 ( Pt 5):643-6. doi: 10.1038/eye.1999.174. PMID 10696317
- [Background] Nischal KC, Khopkar U. Dermoscope. Indian J Dermatol Venereol Leprol. 2005 Jul-Aug;71(4):300-3. doi: 10.4103/0378-6323.16633. No abstract available. PMID 16394450
- [Background] Inui S, Nakajima T, Nakagawa K, Itami S. Clinical significance of dermoscopy in alopecia areata: analysis of 300 cases. Int J Dermatol. 2008 Jul;47(7):688-93. doi: 10.1111/j.1365-4632.2008.03692.x. PMID 18613874